CLINICAL TRIAL: NCT00102024
Title: A Phase I/II, Open-Label, Dose-Escalation Study to Evaluate the Safety and Activity of Single Dose 90Y-Labeled IDEC-159, Humanized, Domain Deleted, Anti TAG-72 Monoclonal Antibody, in Subjects With Metastatic Colorectal Adenocarcinoma
Brief Title: Safety and Activity of 90Y-Labeled IDEC-159 in Subjects With Metastatic Colorectal Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Study MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 159-01
Record Dates: First submitted 2005-01-19; First posted 2005-01-20 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Colorectal Cancer; Metastases
Keywords: Metastatic Colorectal Adenocarcinoma; Anti TAG-72; Monoclonal Antibody
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: Unconjugated IDEC-159
Drug: 111In-IDEC-159
Drug: 90Y-IDEC-159

SUMMARY:
This is a Phase I/II open-label, dose-escalating study in patients with metastatic colorectal cancer. The objectives of the study are to obtain information on the safety of radiolabeled IDEC-159, as well as its activity in colorectal cancer. Another objective is to determine the maximum tolerated dose (MTD). The study duration is 2 years with visits occuring daily and/or weekly for the first 3 months, and every 6 weeks until the end of the 2 year period.

ELIGIBILITY:
Inclusion Criteria:

* Sign an Institutional Review Board (IRB)-approved informed consent.
* Metastatic colorectal adenocarcinoma that has been pathologically confirmed following failed response or relapse while on or following fluoropyrimidine, irinotecan, and oxaliplatin chemotherapy. (Prior therapy with cetuximab is recommended if the tumors are epidermal growth factor receptor [EGFR] positive.)
* Age 18 or above.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Recovered to baseline toxicity from any significant toxicity associated with prior surgery, chemotherapy, biological therapy, or investigational drug.
* Adequate bone marrow reserve (absolute neutrophil count > 1500 cells/mm3, platelet count > 125,000 cells/mm3, hemoglobin concentration ≥ 10 g/dL).
* Radiographically measurable disease (RECIST criteria).
* Life expectancy of at least 3 months.
* Male and female subjects of reproductive potential must agree to follow accepted birth control methods, as determined by the investigator, during treatment and for 12 months after completion of treatment.

Exclusion Criteria:

* Prior radioimmunotherapy.
* Known presence of central nervous system (CNS) metastasis.
* Any lesion > 7.5 cm.
* Total bilirubin > 2.0 mg/dL.
* Total creatinine > 2.0 mg/dL.
* AST and ALT > 2.5 times upper limit of normal (ULN), if metastases to the liver > 5 times ULN.
* Presence of a second primary malignancy requiring active treatment (except for hormonal therapy).
* Serious non-malignant disease or infection that, in the opinion of either the investigator or sponsor, would compromise protocol objectives.
* History of external beam radiation therapy to > 25% of active bone marrow.
* History of bone marrow or stem cell transplant.
* History of granulocyte colony-stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF) therapy within 2 weeks before Study Day 1.
* History of pegylated G-CSF therapy within 4 weeks before Study Day 1.
* History of major surgery, other than diagnostic surgery, within 4 weeks of Study Day 1.
* History of receiving investigational product within 4 weeks before Study Day 1 or long term toxicity from a previous investigational therapy.
* Known history of HIV or AIDS.
* Concurrent systemic corticosteroid therapy or other immunosuppressive agents, unless for the treatment of computed tomography (CT) dye allergy reactions.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To characterize the safety profile and determine the MTD of 90Y-IDEC-159 in subjects with metastatic colorectal cancer.

SECONDARY OUTCOMES:
To evaluate activity; blood, normal organ, and tumor dosimetry; the immunogenicity and pharmacokinetics of 90Y-IDEC-159; and its effect on soluble TAG-72 (sTAG-72) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero, M.D., Principal Investigator — Comprehensive Cancer Center, University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States